CLINICAL TRIAL: NCT04331002
Title: Success of Long-acting Anti-inflammatories After Anterior Cruciate Ligament and Meniscal Injury
Acronym: SLAM
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding Termination
Sponsor: Austin V Stone (Other)
Responsible Party: Sponsor-Investigator, Austin V Stone, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 53136
Record Dates: First submitted 2019-07-27; First posted 2020-04-02 (Actual); Results first posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Tibial Meniscus Injuries; Tibial Meniscus Tears; Tibial Meniscus, Torn; Anterior Cruciate Ligament Tear
Keywords: Knee; Meniscectomy; Meniscus Repair; Anti-inflammatory; Anterior cruciate ligament
MeSH Terms: conditions — Tibial Meniscus Injuries; Anterior Cruciate Ligament Injuries | interventions — Triamcinolone; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: After providing informed consent prior to ACL reconstruction with meniscal involvement, synovial fluid will be collected and assessed for the concentration of pro-inflammatory cytokine interleukin-1alpha (IL-1a). This will be done to identify patients that present with persistent inflammation after surgery that may be at increased risk of cartilage degradation.
  Patients with elevated IL-1a, defined as concentrations > 5 pg/mL, will then be randomized to one of two groups. The threshold of 5 pg/mL was based on our pilot study of 19 patients.
  For those with elevated IL-1a, eight weeks after surgery the knee will be aspirated and one group will receive a single 32 mg Zilretta injection and the other group will receive a 5 mL saline injection.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The knee will be aspirated and one group will receive a single 32 mg Zilretta injection and the other group will receive a 5 mL saline injection. The syringes will be blinded to ensure that both the investigator administering the injection and the patient will be blinded to the group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Experimental (Experimental): The experimental group will receive a single 32 mg Zilretta injection approximately 8 weeks after meniscus surgery.
  Interventions: Drug: Zilretta
- Placebo (Placebo Comparator): The placebo group will receive a single 5 mL injection of normal saline approximately 8 weeks after meniscus surgery.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Zilretta — ZILRETTA is an injectable suspension that delivers 32 mg of triamcinolone acetonide. It is supplied as a single-dose kit containing one vial of ZILRETTA microsphere powder, one vial of 5 mL diluent, and one sterile vial adapter.
  Other Names: Extended release triamcinolone acetonide
  Arms: Experimental
Other: Placebo — 5 mL normal saline
  Other Names: Saline
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if extended-release triamcinolone acetonide treatment alters the progressive changes in bone shape previously demonstrated after anterior cruciate ligament (ACL) reconstruction with partial meniscectomy or meniscal repair.

DETAILED DESCRIPTION:
Anterior cruciate ligament (ACL) injury initiates a biochemical cascade that leads to cartilage degradation and the development of posttraumatic osteoarthritis (PTOA). ACL and acute traumatic meniscus tears have been linked to the development and progression of PTOA. As such, there is an unmet need to identify treatments that may alter the progression of PTOA following ACL meniscus injury. The overarching hypothesis of this project is that intraarticular administration of long-acting anti-inflammatory agents will alter the progression of PTOA following ACL reconstruction.

The current standard of care for patients with combined ACL and meniscus injuries consists of surgical treatment often with a short course of postoperative physical therapy. However, the current mechanically-based standard of care does not address the persistent inflammatory process that promotes cartilage degradation and PTOA progression. The pro-inflammatory stimulation of meniscus cells increases matrix metalloproteinase (MMP) and cytokine activity, and the combination of pro-inflammatory cytokines and compressive loading like what may be seen during sporting and high demand activities further results in degradative enzyme activity and increased production of pro-inflammatory mediators. In this way, the meniscus plays an active role in promoting the cycle of articular cartilage degradation and PTOA progression after ACL reconstruction.

Reducing MMP and cytokine activity after ACL and meniscus injury may alter the progression of PTOA for this at-risk patient population. After ACL injury and reconstruction demonstrate triamcinolone acetonide effectively reduces cartilage degradation, the inflammatory cascade and corresponding cartilage degradation are reinitiated after surgery, hyaluronate treatment 1 week after surgery unsuccessfully mitigates the inflammatory and catabolic processes, and pain and persistent postsurgical cytokine activity at 4 weeks were predictive of inferior knee biomechanics 6 months after surgery. In addition, long-acting agents may provide a greater treatment effect as temporal regulation of cytokine activity may more successfully alter the pro-inflammatory environment than shorter-duration treatments. These results identify that long-acting anti-inflammatory treatment is needed to alter the path of PTOA following meniscus injury and administration 8 weeks after surgery may offer the optimal timing of treatment.

The model whereby femoral shape change and cytokine activity are mediated by a long-acting anti-inflammatory agent (extended-release triamcinolone acetonide) will be tested. Femoral shape changes have been demonstrated after ACL injury and reconstruction, with shape changes in the first 6 months after surgery correlating with subsequent MRI evidence of cartilage degradation and inferior patient-reported outcomes 3 years postoperatively. A Phase 2a, double-blind, placebo-controlled, randomized controlled trial will be performed. The trial will determine if a long-acting anti-inflammatory agent (extended-release triamcinolone acetonide) improves patient-reported outcomes and/or lessens progressive bone shape changes or cartilage breakdown when compared to placebo (saline). Saline was chosen as the placebo as saline has few potential risks and rare adverse events and is the most commonly used placebo treatment option used in knee osteoarthritis research.

ELIGIBILITY:
Inclusion Criteria:

1. Written consent to participate in the study
2. Male or female greater than or equal to 18 years of age and less than 40 years of age
3. Has been consented to undergo arthroscopic ACL reconstruction with partial meniscectomy or meniscal repair
4. Ambulatory and in good general health
5. Willing and able to comply with the study procedures and visit schedules and able to follow verbal and written instructions.
6. Willing to abstain from use of protocol-restricted medications during the study
7. Females and males who have reproductive potential: Must use highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation (10 weeks; 4 to 14 weeks after surgery)
8. Demonstrate persistent inflammation defined as synovial fluid IL-1a concentration greater than or equal to 5 pg/mL at the time of surgery

Exclusion Criteria:

1. Known allergic reactions to components of the extended-release triamcinolone acetonide (Zilretta®)
2. Reactive arthritis, rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis, or arthritis associated with inflammatory bowel disease
3. History of infection in either knee joint
4. Clinical signs and symptoms of active knee infection or crystal disease in either knee within 1 month of Screening
5. Other surgery or arthroscopy of either knee within 6 months of Screening
6. Intraarticular treatment of any joint with any of the following agents within six (6) months of Screening: any corticosteroid preparation or any biologic agent (e.g., platelet rich plasma (PRP) injection, stem cells, prolotherapy, amniotic fluid injection; investigational or marketed).
7. Intraarticular treatment in either knee with hyaluronic acid (investigational or marketed) within 6 months of Screening
8. Parenteral or oral corticosteroids (investigational or marketed) within 3 months of Screening
9. Inhaled, intranasal or topical corticosteroids (investigational or marketed) within 2 weeks of Screening
10. Females who are pregnant or nursing or plan to become pregnant during the study; men whose female partner plans to conceive during the study
11. Radiographic osteoarthritic changes defined as Kellgren-Lawrence grade 2 or greater (as determined by PI from patient's preoperative X-rays)
12. Inability to read and understand English

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2020-08-21 (Actual); Primary Completion 2022-07-11 (Actual); Study Completion 2022-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Austin Stone, MD, PhD, Study Director — University of Kentucky
Locations (1):
- UK Healthcare at Turfland, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Yes
With the participant's approval and as approved by local Institutional Review Boards (IRBs), de-identified biological samples will be stored at the University of Kentucky Orthopedic Biomarker Repository. These samples could be used to research the causes of osteoarthritis after meniscus injury, its complications and other conditions for which individuals with meniscus injuries are at increased risk, and to improve treatment.
  Before sharing biomarker samples, we will ensure that the participant has given previous consent to the sharing of the information or samples. When we confirm that the previously provided consent is still in effect we will remove identifiers such as (e.g., name, medical record number, or date of birth). We will use a secure electronic log to track information shared without releasing the individual participant's identity.
Supporting Information: Study Protocol
Time Frame: Access to individual participant data will be available 1 year after the final study follow-up has been completed, and will be available until 5 years after the final study follow-up has been completed.
Access Criteria: The researchers requesting access to participant information or samples must complete a questionnaire describing why they need information or samples for their research and how they will use the information or samples. The researchers who receive the information or samples will sign an agreement to use the data responsibly.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental | Placebo
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Research cancelled and 0 participants enrolled in Arm 2
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental | Placebo | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1
Height [Number; unit: inches] | 66.96 |  | 66.96
Weight [Number; unit: pounds] | 169.75 |  | 169.75
Body Mass Index [Number; unit: kg/m2] | 26 |  | 26

OUTCOME MEASURES:

1. Primary Outcome: Change in Bone Shape (Baseline to 4 Months)
Description: Using manual segmentation, the volume of the medial femoral condyle will be quantified from 3-Tesla magnetic resonance imaging (MRI) scans performed before and 4 months after the study injection. Medial condyle volume will be expressed as cm3.
Time Frame: Baseline, 4 months
Population: One participant was enrolled in this study. Due to the possibility that the participant could reasonably be identified due to low enrollment, data cannot be presented.
Arm/Group | Experimental | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change in IKDC (Baseline to 4 Months)
Description: The International Knee Documentation Committee (IKDC) scores range from 0-100 with greater scores being indicative of greater self-reported function and reduced pain.
Time Frame: Baseline, 4 months, 1 year, 2 years
Population: as for outcome 1
Arm/Group | Experimental | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change in IKDC (Baseline to 1 Year)
Description: as for outcome 2
Time Frame: Baseline, 4 months, 1 year, 2 years
Population: as for outcome 1
Arm/Group | Experimental | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change in IKDC (Baseline to 2 Years)
Description: as for outcome 2
Time Frame: Baseline, 4 months, 1 year, 2 years
Population: as for outcome 1
Arm/Group | Experimental | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change in KOOS Global (Baseline to 4 Months)
Description: The Knee injury and Osteoarthritis Outcome Score (KOOS) Global scores range from 0-100 with greater scores being indicative of greater self-reported knee function and reduced pain and symptoms.
Time Frame: Baseline, 4 months, 1 year, 2 years
Population: as for outcome 1
Arm/Group | Experimental | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change in KOOSglobal (Baseline to 1 Year)
Description: as for outcome 5
Time Frame: Baseline, 4 months, 1 year, 2 years
Population: as for outcome 1
Arm/Group | Experimental | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change in KOOSglobal (Baseline to 2 Years)
Description: as for outcome 5
Time Frame: Baseline, 4 months, 1 year, 2 years
Population: as for outcome 1
Arm/Group | Experimental | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change in ICOAP (Baseline to 4 Months)
Description: The Intermittent and Constant Osteoarthritis Pain (ICOAP) Score is a valid and reliable tool to assess osteoarthritis-related pain. Scores range from 0 to 100, with greater scores indicating worse pain.
Time Frame: Baseline, 4 months, 1 year, 2 years
Population: as for outcome 1
Arm/Group | Experimental | Placebo
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Change in ICOAP (Baseline to 1 Year)
Description: as for outcome 8
Time Frame: Baseline, 4 months, 1 year, 2 years
Population: as for outcome 1
Arm/Group | Experimental | Placebo
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Change in ICOAP (Baseline to 2 Years)
Description: as for outcome 8
Time Frame: Baseline, 4 months, 1 year, 2 years
Population: as for outcome 1
Arm/Group | Experimental | Placebo
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Change in CTXII (Baseline to 4 Months)
Description: C-terminal cross-linked telopeptides (CTX); CTXII levels measured by ELISA. CTXII is a biomarker of type II collagen breakdown
Time Frame: Baseline, 4 months
Population: as for outcome 1
Arm/Group | Experimental | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Only 1 participant was enrolled in this study. Based on the low enrolment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.
Description: Only 1 participant was enrolled in this study. Based on the low enrolment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.
Arm/Group | Experimental | Placebo
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-16): https://cdn.clinicaltrials.gov/large-docs/02/NCT04331002/Prot_SAP_000.pdf